CLINICAL TRIAL: NCT00976443
Title: Physiologic Effects of High-Dose Gastric Antral Botulinum Toxin Injections
Brief Title: Effects of Gastric Antral Botulinum Toxin Injections in Obese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Topazian, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-000002
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Obesity
Keywords: Obesity; Gastric Emptying; Satiation; Endosonography; Endoscopy; Feeding Behavior
MeSH Terms: conditions — Obesity; Feeding Behavior | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (normal saline) (Placebo Comparator): Gastric injections of normal saline
  Interventions: Drug: Placebo (normal saline)
- BTA 100 U (Active Comparator): Gastric injections of botulinum toxin A, 100 Units
  Interventions: Drug: BTA
- BTA 300 U (Active Comparator): BTA 300 U, gastric injections under EUS guidance
  Interventions: Drug: BTA

INTERVENTIONS:
Drug: BTA — BTA 100 or 300 U, endoscopic ultrasound (EUS) guided injections into gastric antrum
  Other Names: Botox
  Arms: BTA 100 U; BTA 300 U
Drug: Placebo (normal saline) — Placebo (normal saline), gastric injections of normal saline
  Arms: Placebo (normal saline)

SUMMARY:
Obesity is an important public health problem in the United States. The investigators hypothesize that stomach injections of botulinum toxin A (BTA), delivered through an endoscope using endoscopic ultrasound (EUS), may cause delayed gastric emptying, satiation, and reduction in body weight. This protocol is designed to study the effects and safety of gastric BTA injections. Subjects are randomized to receive placebo or one of two different doses of BTA injected into the stomach during one endoscopy, performed via the mouth. Gastric emptying, satiation, symptoms, psychological dimensions of eating behavior, and caloric intake are recorded before and after injections, and subjects are seen in follow-up for 24 weeks.

DETAILED DESCRIPTION:
Additional information regarding study interventions can be obtained by contacting study staff.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 60 years
* BMI ≥ 35 kg /m²
* No history of diabetes, gastric or small bowel surgery, known gastroparesis, prior peptic ulcer, esophagitis, or gastrointestinal stricture.
* Not pregnant or nursing. Women of childbearing potential must have a negative urine pregnancy test within 48 hours prior to each gastric emptying study, and the Botox injection procedure.

Exclusion Criteria:

* Unable or unwilling to provide written informed consent
* ASA Class III or higher
* Chronic upper abdominal pain, nausea, or vomiting
* Allergy to botulinum toxin
* Delayed gastric emptying (abnormal T ½) on baseline scintigraphic gastric emptying test
* Active esophageal, gastric, or duodenal ulceration at time of diagnostic EGD
* Allergic to both penicillins AND quinolones
* Subject has taken warfarin (Coumadin) or clopidogrel (Plavix) in the week preceding EUS

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in body weight between baseline and 16 weeks after BTA injection. | 16 weeks

SECONDARY OUTCOMES:
Change in BMI and waist circumference | 16 weeks
Change in gastric emptying T½ | Baseline to 2 weeks
Change in nutrient drink test maximum tolerated volume (MTV) | 16 weeks
Change in gastrointestinal symptoms over time | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Topazian, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Topazian M, Camilleri M, De La Mora-Levy J, Enders FB, Foxx-Orenstein AE, Levy MJ, Nehra V, Talley NJ. Endoscopic ultrasound-guided gastric botulinum toxin injections in obese subjects: a pilot study. Obes Surg. 2008 Apr;18(4):401-7. doi: 10.1007/s11695-008-9442-x. Epub 2008 Feb 20. PMID 18286347
- [Derived] Topazian M, Camilleri M, Enders FT, Clain JE, Gleeson FC, Levy MJ, Rajan E, Nehra V, Dierkhising RA, Collazo-Clavell ML, Talley NJ, Clark MM. Gastric antral injections of botulinum toxin delay gastric emptying but do not reduce body weight. Clin Gastroenterol Hepatol. 2013 Feb;11(2):145-50.e1. doi: 10.1016/j.cgh.2012.09.029. Epub 2012 Oct 9. PMID 23063681